CLINICAL TRIAL: NCT00214084
Title: Influence of Xanthine Oxidase Inhibition on Vascular Function in Obstructive Sleep Apnea
Brief Title: Vascular Pathophysiology in Obstructive Sleep Apnea
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 2003-085
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Allopurinol

INTERVENTIONS:
Drug: Allopurinol

SUMMARY:
Obstructive sleep apnea (OSA) is a medical problem whose importance is increasing in recognition and awareness. The National Commission on Sleep Disorders estimates that 15 million Americans have OSA, many of whom remain undiagnosed (24). OSA is associated with the development of hypertension and other cardiovascular diseases (1,2). Patients with OSA, like those with congestive heart failure, hypertension, hypercholesterolemia and diabetes, exhibit impaired EDV (25-32). OSA is also associated with impairments in endothelium-dependent cerebral blood flow responses, which may be a risk factor for stroke (33). Impaired EDV is a result of reduced production or inadequate action of nitric oxide. Since EDV worsens with disease progression and improves with disease treatment, it serves as a prognostic marker of vascular function (34-37). In OSA, hypoxia and neurohumoral disturbances increase generation of reactive oxygen species (ROS) that neutralize nitric oxide and impair endothelium-dependent responses (9,10,38). One source of ROS in endothelial cells is the enzyme xanthine oxidase (38). XO is an enzyme present in the vascular endothelium that significantly contributes to generation of ROS in congestive heart failure, hypercholesterolemia and diabetes (13-17). Inhibition of XO improves endothelium-dependent resistance vessel responses in these populations (13-17), but it is unknown if XO significantly contributes to oxidative stress and endothelial dysfunction in OSA. The central hypothesis of this application is that inhibition of XO with allopurinol will reduce oxidative stress and generation of ROS, thereby improving nitric oxide bioavailability and EDV in OSA. Our hypothesis has been formulated on the basis that patients with OSA experience repeated hypoxemia that increases activity of XO and other enzymes, thus increasing the generation of ROS that negatively impact EDV. Hypoxia is detrimental to vascular homeostasis since it increases generation of ROS through direct mechanisms and via activation of XO.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Sleep Disordered Breathing:
* Significant obstructive sleep apnea as verified by complete overnight polysomnography with apnea-hypopnea index (AHI) > 10 events per hour.
* Fasting total cholesterol < 240 mg/dL
* Fasting blood glucose < 120 mg/dL
* Control subjects:
* Free of sleep disordered breathing verified by complete overnight polysomnography or oxygen desaturation screening (AHI < 5 events per hour)
* Fasting total cholesterol < 240 mg/dL
* Fasting blood glucose < 120 mg/dL

Exclusion Criteria:

* Presence of any cardiovascular diseases or medical conditions that will affect vascular responses (other than sleep apnea)
* Subject taking any vasoactive medications, willing to stop taking vitamins or supplements for study participation
* Current smokers
* History of adverse reaction to allopurinol, acetylcholine, nitroprusside, verapamil or lidocaine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Forearm resistance ratios between the infused and non-infused arms at the highest dose of acetylcholine (30 mcg/minute)

SECONDARY OUTCOMES:
Area under the curve in reduction of forearm resistance during acetylcholine following allopurinol compared to placebo

CONTACTS AND LOCATIONS:
Overall Officials: John M Dopp, PharmD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States